CLINICAL TRIAL: NCT03821610
Title: A Comparison of Reduced Dose Total Body Irradiation (TBI) and Cyclophosphamide With Fludarabine and Melphalan Reduced Intensity Conditioning in Adults With Acute Lymphoblastic Leukaemia (ALL) in Complete Remission. (ALL-RIC)
Acronym: ALL-RIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-241
Record Dates: First submitted 2019-01-09; First posted 2019-01-30 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Melphalan; Alemtuzumab; Cyclophosphamide; Mesna; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fludarabine / Melphalan / Alemtuzumab (Active Comparator): Day -7 Fludarabine 30mg/m2 od IV Day -6 Fludarabine 30mg/m2 od IV Day -5 Fludarabine 30mg/m2 od IV Day -4 Fludarabine 30mg/m2 od IV Day -3 Fludarabine 30mg/m2 od IV Day -2 Melphalan 140mg/m2 od IV, Alemtuzumab 20 mg od IV (unrelated transplants only) Day -1 Alemtuzumab 20mg od IV Day 0 Infusion of sibling or unrelated donor peripheral blood stem cells
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Alemtuzumab
- Cyclophosphamide / TBI (8Gy) (Experimental): Day -6 Cyclophosphamide 50 mg/kg od IV , Mesna 20 mg/kg od IV, Mesna 76mg/kg od IV Day -5 Cyclophosphamide 50 mg/kg od IV, Mesna 20 mg/kg od IV, Mesna 76 mg/kg od IV Day -4 Rest Day -3 TBI (2Gy) bd Day -2 TBI (2Gy) bd, Alemtuzumab 20mg od IV (unrelated transplants only) Day -1 Alemtuzumab 20mg od IV Day 0 Infusion of sibling or unrelated donor peripheral blood stem cells or bone marrow
  Interventions: Drug: Alemtuzumab; Drug: Cyclophosphamide; Drug: Mesna; Radiation: Total Body Irradiation (8Gy)

INTERVENTIONS:
Drug: Fludarabine — IV
  Arms: Fludarabine / Melphalan / Alemtuzumab
Drug: Melphalan — IV
  Arms: Fludarabine / Melphalan / Alemtuzumab
Drug: Alemtuzumab — IV
Drug: Cyclophosphamide — IV
  Arms: Cyclophosphamide / TBI (8Gy)
Drug: Mesna — IV
  Arms: Cyclophosphamide / TBI (8Gy)
Radiation: Total Body Irradiation (8Gy) — TBI (8Gy)
  Arms: Cyclophosphamide / TBI (8Gy)

SUMMARY:
The current national acute lymphoblastic leukaemia (ALL) trial in adults investigated whether a low (reduced) intensity chemotherapy regimen prior to transplant could improve the outcome of patients with ALL who are over 40 years of age. The results (60% 2 year survival) are very encouraging but patients who come to transplant with small amounts of 'residual' disease had less good outcomes. The goal of this trial is to see if a slightly stronger chemotherapy regimen (involving total body irradiation, (TBI)) can improve results by reducing the chance of the disease coming back (relapsing) without increasing the chance of not surviving the transplant. Up to 242 patients will be 'randomised' to the trial to receive either the established chemotherapy of fludarabine and melphalan or cyclophosphamide and TBI to compare the outcomes between the two treatment regimens. Other measures to reduce relapse will be the earlier use of donor white cell infusions and earlier stopping of immune suppressive drugs to enhance the immune effect of the transplanted cells (graft). Patients will be followed up for a minimum of 3 years. All patients on the next national ALL trial (UKALL XV) will be offered this trial but it will also be open to patients not on this study.

DETAILED DESCRIPTION:
TRIAL SYNOPSIS

Trial Design This is a 2 arm, phase II, multicentre, randomised clinical trial in adult patients with ALL in complete remission (CR) undergoing allogeneic stem cell transplantation (SCT) comparing the novel conditioning regimen of TBI and cyclophosphamide with the standard condition of Fludarabine/Melphalan/Alemtuzumab (FMA).

Patient will be stratified at randomisation by the donor type (sibling; suitable matched), CR status (CR1; CR2) and by age (above; below 55 years of age). Patients eligible for entry into the trial will be randomised on a 1:1 basis to receive either the experimental treatment arm or the control arm.

Objectives Primary Objectives To compare the disease free survival (DFS) at two years of patients with ALL after a TBI and cyclophosphamide allograft with that of patients transplanted using the FMA conditioning regimen.

Secondary Objectives To compare overall survival (OS), cumulative incidence of disease relapse (CIR), non-relapse mortality (NRM), incidence of grade 2-4 acute graft-versus-host-disease (GvHD), incidence of chronic GvHD of any grade, occurrence and severity of veno-occlusive disease (VOD), duration of hospitalisation in the first year, quality of life (QoL), full donor chimerism at day 100 and TBI related symptomatic pulmonary toxicity between the control and experimental arm following allogenic SCT.

Exploratory Objectives To measure multi-lineage chimerism and molecular minimal residual disease (MRD) at 3 monthly intervals and the ability of planned donor lymphocyte infusion (DLI) to 'correct' mixed chimerism and reverse molecular relapse/persistence and reduce the incidence of frank haematologic relapse.

To ascertain if either of the conditioning arms is more effective in controlling disease in patients who are MRD positive before transplant.

Patient Population This trial will recruit patients with ALL in CR as defined by the WHO classification (Appendix 1). Patients enrolled onto the UKALL XIV registration study and the planned national UKALL XV study who are eligible for transplant will also be able to enrol onto ALL-RIC provided they meet the entry criteria.

Sample Size A minimum of 247 patients will be randomised 1:1 between the control and experimental treatment arms.

Trial Duration Patients will be recruited over 48 months across IMPACT centres. Patients will be followed up for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40-70 years. NB: Patients under the age of 40 who are considered unsuitable for a myeloablative transplant may enrol onto the trial following discussion with the CI via the Trials Office
* Patients with ALL in first or second CR
* Availability of a human leukocyte antigen (HLA) identical sibling or suitable matched donor (suitable matched defined as no greater than a single allele mismatch at HLA A, B, C or DRβ1). A single allele mismatch is permitted if there are adverse cytogenetics or MRD positivity at any timepoint
* Patients considered suitable to undergo a RIC allogeneic SCT as clinically judged by the Local Investigator including:-

  * Adequate hepatic and renal function as determined by full blood count and biochemistry assessment
  * Resolution of any toxic effects of prior therapy (including radiotherapy, chemotherapy or surgical procedures). Patients with bone marrow suppression following therapy may enter the trial
  * Patients with abnormal cardiac and/or pulmonary function must be considered fit for allogeneic SCT including 8Gy of TBI at the time of randomisation.
* Patients with an ECOG performance status 0,1 or 2
* Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must use appropriate, highly effective, contraception from the point of admission for transplant conditioning therapy until 12 months after transplant (see section 8.1.2.2)
* Patients have given written informed consent
* Patients willing and able to comply with scheduled study visits and laboratory tests

Exclusion Criteria:

* Patients with contraindications to receiving RIC allogeneic SCT
* Female patients who are pregnant or breastfeeding. All women of childbearing potential (WOCBP) must have a negative pregnancy test before commencing treatment
* Adults of reproductive potential not willing to use appropriate, effective, contraception during the specified period
* Patients with renal or hepatic impairment as clinically judged by Local Investigator
* Patients with active infection, HIV-positive or chronic active Hep-A or -C
* Patients with concurrent active malignancy. Patients with a previous history of malignancy can be included if that malignancy is considered to be at a low risk of recurrence
* Previous exposure to a high dose of radiotherapy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | The main analysis will take place once all patients have completed 2 years of follow up.
  Defined as time from randomisation to the first of relapse or death from any cause. Patients who are still alive and progression free at the end of the trial will be censored at their last date known to be alive.

SECONDARY OUTCOMES:
Overall Survival (OS) | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
  Defined as time from randomisation to date of death from any cause. Patients who are alive at the end of the trial will be censored at their date last known to be alive
Cumulative Incidence of Relapse (CIR) | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
  Defined as time from randomisation to the date of relapse. Patients who die without relapse will be treated as a competing risk and patients who are alive and relapse free at the end of the trial will be censored as their date last seen
Non-relapse mortality (NRM) | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
  Defined as time from randomisation to death from any cause that occurred without relapse. Patients who relapse will be treated as a competing risk and patients who are still alive and relapse free at the end of the trial will be censored at their date last known to be aliveIncidence of Grade 2-4 acute GvHD within 100 days of transplant
Incidence of chronic GvHD of any grade at 2 years | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
Occurrence and severity of VOD (Veno-occlusive disease) in the first 100 days | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
Duration of hospitalisation | The outcome will be conducted when all patients have completed 1 year of follow up.
  Duration of hospitalisation recorded between start of conditioning regimen and 1 year post transplantation.
Quality of Life (QoL) assessment (FACT-BMT Questionnaire) | Collected at baseline, Day 100, Month 12, Month 24, Month 36, Month 48 and Month 60 for each patient. The outcome will be analysed when the last patient has completed 2 years of follow up.
  FACT-BMT Questionnaire uses Units on a scale 0-4. It measures quality of life, with 0 being the lowest quality of life and 4 being the highest quality of life.
Quality of Life (QoL) assessment (Short Form 36 Health Survey) | Collected at baseline, Day 100, Month 12, Month 24, Month 36, Month 48 and Month 60 for each patient. The outcome will be analysed when the last patient has completed 2 years of follow up.
  Short Form 36 Health Survey uses Units on a scale 1-6. Question 1 & 2 consider general health (1 = best health score, 5 = worst). Question 3 considers activity level (1= least active, 3 = most). Question 4/5 considers work (1= work affected, 2= work not affected). Question 6 considers quality of relationships (1=not affected, 5 = most affected). Question 7 considers pain (1= no pain, 6 = worst). Question 8 considers housework/ paid work (1= not affected, 5= most affected). Question 9 considers mental health (1= best mental health, 6= worst). Question 10 considers social activities (1=most affected, 5= least affected). Question 11 considers self perception (1= worst, 5= best)
Full donor chimerism | The outcome will be analysed when all patients have completed 100 days follow up.
  Number of patients with full donor chimerism at day 100 Follow Up (for each patient)
Occurrence and severity of TBI related symptomatic pulmonary toxicity | Collected in first 12 months from start of treatment
  Collected using CTCAE 4.0 criteria

OTHER OUTCOMES:
Correlation of multi-lineage chimerism and relapse | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up
Correlation of Minimal Residual Disease (MRD) with relapse | The main analysis will take place once all patients have completed 2 years of follow up. A subsequent analysis of long terms outcomes will be completed when all patients have completed 5 years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: David Marks, Study Chair — Bristol Haeamatology and Oncology Centre
Locations (22):
- United Kingdom (22):
  - Heart of England Nhs Foundation Trust, Birmingham
  - University Hospitals Birmingham Nhs Foundation Trust, Birmingham
  - University Hospitals Bristol Nhs Foundation Trust, Bristol
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals Nhs Trust, Leeds
  - University Hospitals of Leicester Nhs Trust, Leicester
  - The Clatterbridge Cancer Centre Nhs Foundation Trust, Liverpool
  - Barts Health Nhs Trust, London
  - University College London Hospitals Nhs Foundation Trust, London
  - Kings College Hospital, London
  - The Royal Marsden Nhs Foundation Trust, London
  - Imperial College Healthcare Nhs Trust, London
  - The Christie Nhs Foundation Trust, Manchester
  - Central Manchester University Hospitals Nhs Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Oxford University Hospitals Nhs Foundation Trust, Oxford
  - Plymouth Hospitals Nhs Trust, Plymouth
  - Sheffield Teaching Hospitals Nhs Foundation Trust, Sheffield
  - University Hospital Southampton Nhs Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No